CLINICAL TRIAL: NCT01029275
Title: Multicenter, Randomised Open Trial Comparing the Efficacy of a Medical Treatment With Sandostatin LP 30 mg Performed Before Surgery to a Prime Line transsphenoïdal Surgery in Previously Untreated Acromegalic Patients With Either a Micro or a Macro Pituitary Adenoma
Brief Title: Somatostatin Analog Treatment of Acromegaly Before Pituitary Surgery : Comparison With Neurosurgery Alone
Acronym: SAPORO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2004/089/HP; 2004-004524-12 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Acromegaly
Keywords: Acromegaly; pituitary adenoma; octreotide; transsphenoïdal surgery; GH; IGF-1
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): pre-operative medical treatment with Sandostatin
  Interventions: Drug: Pre-treatment with octreotide
- Arm B (No Intervention): pituitary surgery as a first line treatment

INTERVENTIONS:
Drug: Pre-treatment with octreotide — Pre-treatment with octreotide
  Arms: Arm A

SUMMARY:
The aim of the study is to evaluate the interest of a six month pre-operative treatment with a long-acting somatostatin analog (Sandostatin LP) versus surgery alone in patients with a pituitary adenoma responsible for acromegaly.

DETAILED DESCRIPTION:
Somatotroph pituitary adenoma is the most frequent cause of acromegaly. A transsphenoidal removal of the tumor is used as the first line treatment. Somatostatin analogs are used as to whether recovery was not obtained after surgery or pituitary surgery was contraindicated. Previous studies with somatostatin analogs have shown a drop in plasma GH and IGF-1 levels and a reduction in adenoma size in 75 and 25% of patients respectively. Retrospective studies suggest that a treatment with somatostatin analogs performed before surgery may be of interest to improve anesthesic conditions and surgical outcome. The aim of present study is to prospectively evaluate the interest of a first line treatment with a long-acting somatostatin analog (Sandostatin) before performing a pituitary surgery in acromegalic patients with either a micro or a macroadenoma to improve peri-operative conditions and hopefully surgical outcome. After informed consent, untreated acromegalic patients will be included and randomly assigned to one of the following treatment procedures : either pituitary surgery or a six month treatment with long-acting Sandostatin 30 mg monthly for 6 months before performing transsphenoïdal adenoma removal. The patients will be evaluated before any treatment, on months 3 and 6 of the treatment with Sandostatin (for the patients enrolled in this arm of the study) and on months 3 and 12 after pituitary neurosurgery. Each evaluation will include clinical data, hormone testing and radiological (MRI) investigation. The main endpoint will be the rate of recovery proved by a normalisation of GH secretion and plasma IGF-1 level. Secondary endpoints will include the evaluation of clinical, radiological, biological, anesthesic, surgical and pathological parameters. A comparison between the two arms will be performed at entry into the study, at the time of surgery and then on months 3 and 12 following the transsphenoidal removal of the somatotroph adenoma.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* 18-80 years old
* untreated acromegaly
* unsuppressed GH secretion after a glucose load and elevated IGF-1 plasma levels
* presence of a pituitary adenoma on MRI
* informed consent given.

Exclusion Criteria:

* acromegaly previously treated
* contraindication to pituitary surgery
* associated hyperprolactinemia above 200 ng/ml
* visual field defect needing rapid transsphenoidal surgery
* contraindication to a treatment with octreotide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
IGF1 plasma levels | 3 months and 12 months after transphenoidal surgery

SECONDARY OUTCOMES:
GH plasma levels | 3 and 12 months after transphenoidal surgery
Evaluation of the effects of the pre-operative treatment with Sandostatin on clinical, radiological, biological, anesthesic, surgical and pathological parameters. | at transphenoidal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Kuhn, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (13):
- France (13):
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Caen University Hospital, Caen
  - Grenoble University Hospital, Grenoble
  - Paris XI University Hospital, Le Kremlin-Bicêtre
  - Lille University Hospital, Lille
  - University Hospital of Limoges, Limoges
  - Lyon University Hospital, Lyon
  - Marseille University Hospital, Marseille
  - Bordeaux University Hospital, Pessac
  - Rouen University Hospital, Rouen
  - Strasbourg University Hospital, Strasbourg
  - Toulouse Universtiy Hospital, Toulouse